CLINICAL TRIAL: NCT06547112
Title: A Pharmacodynamic Study of the Apheresis Product of Multiple Myeloma Patients Undergoing Quad-induction Followed by Motixafortide + G-CSF Mobilization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: BioLineRx, Ltd. (Industry); Arvrmid Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202408102
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Hematopoietic stem cell mobilization; CXCR4 inhibition; Motixafortide; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 4-fluorobenzoyl-TN-14003; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: The study will comprise 2 cohorts enrolled sequentially, each with 10 subjects. The first 10 patients will be enrolled to Cohort 1, and the next 10 patients will be enrolled to Cohort 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Standard dosing (Active Comparator): For Cohort 1, motixafortide will be given on Day 4 between 6:00 and 8:00 pm. A second dose may be given on Day 6 between 6:00 and 8:00 p.m. if CD34+ cell collection goals are not met on Day 5 apheresis.
  Interventions: Drug: Motixafortide; Drug: G-CSF
- Cohort 2: Early dosing (Experimental): For Cohort 2, motixafortide will be given on Day 4 between 2:00 and 4:00 pm. A second dose may be given on Day 6 with goal of administration between 6:00 and 8:00 pm after completion of pheresis if clinically feasible. if CD34+ cell collection goals are not met on Day 5 apheresis.
  Interventions: Drug: Motixafortide; Drug: G-CSF

INTERVENTIONS:
Drug: Motixafortide — Dose = 1.25 mg/kg via subcutaneous injection
  Other Names: BL-8040
Drug: G-CSF — Dose = ~10 µg/kg (and maximum of 15 µg/kg) via subcutaneous injection

SUMMARY:
This study includes extended CD34+ profiling on the apheresis product of multiple myeloma patients undergoing standard-of-care quad-induction followed by motixafortide + G-CSF mobilization, and in addition, assesses the pharmacodynamics (PD) of motixafortide following "standard" (~12 hours) vs "early" (~16 hours) dosing. The investigators hypothesize that quad-induction may alter the stem cell subsets within the mobilized graft. The investigators further hypothesize that standard and early dosing strategies will result in comparable mobilization and stem cell collection rates.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 18 and 78 years, inclusive.
* Histologically confirmed multiple myeloma expected to receive high-dose chemotherapy (HDT) and autologous stem cell transplantation (ASCT)
* Received ≥3 cycles but ≤6 cycles of daratumumab-based quadruplet induction therapy (quadruplet induction therapy: combining daratumumab, a proteasome inhibitor, an IMiD, and dexamethasone) before ASCT
* At least one week (7 days) from last induction cycle prior to the first dose of G-CSF for mobilization
* The subjects should be in first or second CR (including CR and SCR) or PR (including PR and VGPR)
* ECOG performance status 0 or 1
* Adequate organ function at screening as defined below:

  * White blood cell (WBC) counts > 2.5 × 10^9/L
  * Absolute neutrophil count > 1.5 K/cumm
  * Platelet count >100 K/cumm
  * GFR value of ≥15 mL/min/1.732 (by MDRD equation)
  * ALT and/or AST ≤2.5 × ULN
  * Total bilirubin ≤2.0 × ULN unless the participant has Gilbert disease
  * INR or PT: ≤1.5 × ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT: ≤1.5 × ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Female subjects must be of non-childbearing potential or, if of childbearing potential, must have a negative serum pregnancy test at screening and negative urine or serum pregnancy test within 7 days prior to G-CSF first administration.

Non-childbearing potential is defined as (by other than medical reasons):

* ≥45 years of age and has not had menses for over 2 years
* Post hysterectomy, bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation at least 6 weeks prior to screening

  * Women of childbearing potential must agree to use 2 methods of effective contraception: One barrier method (e.g., diaphragm, or condom or sponge, each of which are to be combined with a spermicide) and one hormonal method, unless she uses a highly effective method. Highly effective methods of contraception include:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable, intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized partner
* Sexual abstinence These methods must be used starting at study enrollment and for the duration of study participation through 8 days after the last dose of motixafortide.

Male subjects must agree to use an adequate method of contraception (barrier method) starting with the first day of G-CSF administration through 8 days after the last dose of motixafortide.

* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Previous history of autologous or allogeneic-HCT
* Failed previous HSC collections or collection attempts
* Taken any of the listed below concomitant medications, growth factors or stimulating agents within the designated washout period:

  * Dexamethasone: 7 days
  * Thalidomide: 7 days
  * Lenalidomide: 7 days
  * Pomalidomide: 7 days
  * Bortezomib: 7 days
  * Carfilzomib: 7 days
  * Ixazomib: 7 days
  * G-CSF: 14 days
  * GM-CSF or pegfilgrastim: 21 days
  * Erythropoietin or erythrocyte-stimulating agents: 30 days
  * Eltrombopag, romiplostim or platelet-stimulating agents: 30 days
  * Carmustine (BCNU): 42 days/6 weeks
* Received >6 cycles lifetime exposure to an IMiD
* Received >8 cycles of alkylating agent combinations
* Received >6 cycles of melphalan
* Received prior treatment with radioimmunotherapy (e.g., radionuclides, holmium)
* Received prior treatment with venetoclax
* Has received a live vaccine within 30 days of the planned start of G-CSF administration. Seasonal flu vaccines that do not contain live virus are permitted.
* Known active CNS metastases or carcinomatous meningitis
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to motixafortide, G-CSF or other agents used in the study
* Has an active or uncontrolled infection requiring systemic therapy
* Has a known additional malignancy that is progressing or requires active treatment
* Has a known underlying medical condition that, in the opinion of the treating physician or Principal Investigator, would preclude study participation.
* Is currently participating in an investigational treatment study, or has participated in a study of an investigational agent and received study therapy, or has been treated with an investigational device, within 4 weeks prior to the first dose of treatment.
* O2 saturation < 92% (on room air)
* Personal history or family history of long QT syndrome or torsade de pointes
* History of unexplained syncope, syncope from an uncorrected cardiac etiology, or family history of sudden cardiac death.
* History of myocardial infarction, CABG, coronary or cerebral artery stenting and/or angioplasty, stroke, cardiac surgery, or hospitalization for congestive heart failure within 3 months prior to study enrollment, Angina Pectoris Class >2 or NYHA Heart Failure Class >2.
* ECG at screening showing QTcF >470 msec and/or PR >280 msec
* Mobitz II 2nd degree AV Block, 2:1 AV Block, High Grade AV Block, or Complete Heart Block, unless the participant has an implanted pacemaker or implantable cardiac defibrillator (ICD) with backup pacing capabilities.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the treating physician or Principal Investigator.
* Is pregnant or breast-feeding or expecting to conceive or women of childbearing potential unless consent to use two contraceptive methods or highly effective contraception as detailed above, within the projected duration of the trial, starting with the Screening Visit through 8 days after the last dose of study drug.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Absolute number and relative proportions of CD34+ cell subsets by extended immunophenotypic profiling using multicolor fluorescence activated cell sorting (mFACS) on the apheresis product | From day 5 through day 8 (up to 4 days)

SECONDARY OUTCOMES:
Number of participants with adverse events | From day 4 to end of study visit (estimated to be 15-26 days)
Change in concomitant medication use | From baseline through end of study visit (estimated to be 15-26 days)
Treatment compliance | From day 4 to end of study visit (estimated to be 15-26 days)
Number of participants who dropout due to adverse events | From day 4 to end of study visit (estimated to be 15-26 days)
Change in blood pressure | From baseline through end of study visit (estimated to be 15-26 days)
Change in temperature | From baseline through end of study visit (estimated to be 15-26 days)
Change in heart rate | From baseline through end of study visit (estimated to be 15-26 days)
Change in respiratory rate | From baseline through end of study visit (estimated to be 15-26 days)
Change in oxygen saturation at room air | From baseline through end of study visit (estimated to be 15-26 days)
Kinetics of PD assessed by the number of CD34+ cells/μL in peripheral blood | 0, +2, +4, +8, + 12 hours in Cohorts 1 and 2, +16 hours in Cohort 2, and, if needed +36 hours in Cohort 1 or +40 hours in Cohort 2
Apheresis yields assessed by total CD34+ cells/kg in apheresis product | At 12 hours in Cohort 1 and 16 hours in Cohort 2
Proportion of participants who mobilize ≥2.0 × 10^6 CD34+ cells/kg | In up to 2 apheresis sessions - from day 5 through day 8 (up to 4 days)
Proportion of participants who mobilize ≥5.0 × 10^6 CD34+ cells/kg | In up to 2 apheresis sessions - from day 5 through day 8 (up to 4 days)
Proportion of participants who mobilize ≥6.0 × 10^6 CD34+ cells/kg | In up to 2 apheresis sessions - from day 5 through day 8 (up to 4 days)
Proportion of participants who mobilize ≥2.0 × 10^6 CD34+ cells/kg | In up to 1 apheresis session - from day 5 through day 8 (up to 4 days)
Proportion of participants who mobilize ≥5.0 × 10^6 CD34+ cells/kg | In up to 1 apheresis session - from day 5 through day 8 (up to 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Crees, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu